CLINICAL TRIAL: NCT02265081
Title: A Prospective Study on USS Assessment of Pelvic Structures in 3rd Trimester of Pregnancy Versus Delivery Outcome.
Acronym: PLUSSMODEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birmingham Women's NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Aneta Obloza, DR ANETA OBLOZA, Birmingham Women's NHS Foundation Trust
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: U1111-1162-7720
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Pelvic Floor Disorders; Pregnancy
MeSH Terms: conditions — Pelvic Floor Disorders | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- nulliparous women (Active Comparator): internal ultrasound in the 3rd trimester uroflow meter in 3rd trimester
  Interventions: Procedure: ultrasound; Procedure: uroflow-meter
- parous women (Experimental): those who had vaginal delivery in the past; internal ultrasound in the 3rd trimester uroflow meter in 3rd trimester
  Interventions: Procedure: ultrasound; Procedure: uroflow-meter
- parous women - VBAC (Experimental): those with previous LSCS and no vaginal births; internal ultrasound in the 3rd trimester uroflow meter in 3rd trimester
  Interventions: Procedure: ultrasound; Procedure: uroflow-meter

INTERVENTIONS:
Procedure: ultrasound — pelvic floor ultrasound
Procedure: uroflow-meter — uroflow meter: measurement of passed urine volume

SUMMARY:
The proposed study is to evaluate if there are specific factors in the pelvic floor functional anatomy which can predict the ability of having a vaginal birth after caesarean section.

Physical characteristics of the soft tissue in the female pelvis play an important role in successful vaginal delivery. A "tight" or less distensible pelvic floor muscles may influence mode of delivery, leading to poor labour progression and by compressing foetal head produce CTG abnormality such as decelerations, both resulting in caesarean delivery.

One of the main structures of the pelvic floor, the puborectoalis muscle, facilitates the passage of fetal head through the birth canal by stretching and distending. Therefore distensibility of the female pelvic floor influences mode of delivery.

Three hundred patients, in the third trimester of pregnancy, will be recruited via the antenatal clinics to minimize any disruption in their pregnancy care provision. Eligible participants are pregnant women who had either one or no vaginal births, or one caesarean section and who can give an informed consent and maintain their autonomy regarding mode of delivery with understanding of the forthcoming study results. Participants will be excluded if they sustain any obstetric complications that may impede on time and mode of delivery including an emergency prelabour caesarean section.

Ultrasonographic assessment of the differences in the pelvic characteristics of these women will be used to predict a successful of trial of vaginal delivery after caesarean section (VBAC) in subsequent pregnancies. The results will be used to better inform whether there is a simple (single ultrasound assessment) that can be used to help inform women's choice regarding mode of delivery.

Results from this research could be a pioneering blueprint for further studies, as there is very little known about this topic.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking women
2. over 16 years old women
3. women willing to provide written informed consent
4. women who had either prior vaginal delivery or caesarean section or no prior birth experience

Exclusion Criteria:

1. Women who cannot give an informed consent,
2. under the age of consent,
3. any participants whose pregnancies complicated during the antenatal period that may influence decision on time and mode of delivery that is anyone who has to undergo an emergency prelabour LSCS,
4. nonEnglish speaking women
5. less than 16 years old women

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 135 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
vaginal delivery | 12 months

SECONDARY OUTCOMES:
voiding problems | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Hard, Study Chair — R&D Dept, Birmingham Women's Hospital, UK
Locations (1):
- Birmingham Women's Hospital, Birmingham, United Kingdom